CLINICAL TRIAL: NCT05223062
Title: Self-Reported Medication Adherence in Patients With Psoriatic Arthritis: Influence of Illness Perception and Medication Beliefs
Brief Title: Medication Adherence in Psoriatic Arthritis
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/263
Record Dates: First submitted 2022-01-23; First posted 2022-02-03 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic Arthritis; Medication Adherence
MeSH Terms: conditions — Arthritis, Psoriatic; Medication Adherence | interventions — 4-amino-4'-hydroxylaminodiphenylsulfone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Psoriatic arthritis: Patients with psoriatic arthritis according to the Classification Criteria for Psoriatic Arthritis (CASPAR).
  Interventions: Other: Disease activity in psoriatic arthritis (DAPSA); Other: Compliance-Questionnaire-Rheumatology (CQR); Other: The Brief Illness Perception Questionnaire (BIPQ); Other: The Beliefs About Medicines Questionnaire (BMQ); Other: Hospital Anxiety and Depression Scale (HADS); Other: The Psoriatic Arthritis Quality of Life (PsAQoL)

INTERVENTIONS:
Other: Disease activity in psoriatic arthritis (DAPSA) — DAPSA includes a 68/66 joint count summed with a patient global, patient pain score, and C- reactive protein level. The DAPSA provides a continuous score of arthritis activity and has validated cut points for remission (< 4) and low disease activity (< 14).
Other: Compliance-Questionnaire-Rheumatology (CQR) — The CQR is a self-administered questionnaire that was developed with the aim of correctly identifying patients that were classified as "low" adherers (taking <80% of their medication correctly). The four point Likert answering scale ranges from; "Definitely don't agree" (scored 1) to "Definitely agree" (scored 4) with lower scores indicating lower levels of adherence. Total score is between 0 and 100.
Other: The Brief Illness Perception Questionnaire (BIPQ) — The Brief Illness Perception Questionnaire (BIPQ) is a questionnaire that assesses a number of beliefs about illness which are thought to be related to coping and help-seeking behavior. Each item is scored between 0 and 10. Maximum total score is 80. Higher scores represents that the patient has a concerned perception of illness.
Other: The Beliefs About Medicines Questionnaire (BMQ) — The Beliefs About Medicines Questionnaire (BMQ) is a tool for evaluating people's beliefs about medicines. The BMQ comprises two sections: the BMQ-Specific which assesses representations of medication prescribed for personal use and the BMQ-General which assesses beliefs about medicines in general. It has a total of 18 questions scored with a 5-point Likert scale. Higher scores represent more powerful beliefs.
Other: Hospital Anxiety and Depression Scale (HADS) — Hospital Anxiety and Depression Scale (HADS) determines the levels of anxiety and depression that a person is experiencing. The HADS is a fourteen item scale that generates: Seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression.
Other: The Psoriatic Arthritis Quality of Life (PsAQoL) — The Psoriatic Arthritis Quality of Life (PsAQoL) measure is a disease specific patient-reported outcome measure which measures the effect that psoriatic arthritis has on a patient's quality of life. It is a self-administered, 20-item questionnaire that takes about three minutes to complete. The answers are restricted to true or false.A high score on the PsAQoL indicates a lower quality of life. Total score is between 0 and 20.

SUMMARY:
Psoriatic arthritis (PsA) is a chronic multisystemic disease requiring ordinary doctor visits and an adherence to medication. Evaluating the parameters affecting the medication adherence is essential for the efficacy of the treatment. To our knowledge no study has ever evaluated the factors affecting the medication adherence in patients with PsA so far.

DETAILED DESCRIPTION:
Psoriatic arthritis (PsA) is a multisystemic disease requiring ordinary doctor visits and an adherence to medication. Due to its chronic nature treatment regimens lasts for the lifetime and that may affect the efficacy of the treatment. Although treatment with drugs is a biological intervention, medication adherence and eliminating the factors affecting it seems essential for treatment efficacy. To our knowledge no study has ever evaluated the factors affecting the medication adherence in patients with PsA so far. Our aim in this study is to evaluate the factors affecting the medication adherence in patients with PsA.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with PsA according to CASPAR criteria
* Administering PsA medication for at least 6 moths
* Aged ≥18

Exclusion Criteria:

* Not having enough cognitive functions to understand and answer the questionnaires
* Having a psychiatric disorder
* Having a severe comorbidity (e.g. malignancy, stroke)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with psoriatic arthritis having medication for at least 6 months
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Disease activity in psoriatic arthritis (DAPSA) | 1 day
  The score of Disease activity in psoriatic arthritis (DAPSA) provides a continuous score of arthritis activity and has validated cut points for remission (< 4) and low disease activity (< 14). Higher scores represent a worse outcome.
Compliance-Questionnaire-Rheumatology (CQR) | 1 day
  The CQR is a self-administered questionnaire that was developed with the aim of correctly identifying patients that were classified as "low" adherers (taking <80% of their medication correctly). The four point Likert answering scale ranges from; "Definitely don't agree" (scored 1) to "Definitely agree" (scored 4) with lower scores indicating lower levels of adherence. Total score is between 0 and 100.
The Brief Illness Perception Questionnaire (BIPQ) | 1 day
  The Brief Illness Perception Questionnaire (BIPQ) is a questionnaire that assesses a number of beliefs about illness which are thought to be related to coping and help-seeking behavior. Each item is scored between 0 and 10. Maximum total score is 80. Higher scores represents that the patient has a concerned perception of illness.
The Beliefs About Medicines Questionnaire (BMQ) | 1 day
  he Beliefs About Medicines Questionnaire (BMQ) is a tool for evaluating people's beliefs about medicines. The BMQ comprises two sections: the BMQ-Specific which assesses representations of medication prescribed for personal use and the BMQ-General which assesses beliefs about medicines in general. It has a total of 18 questions scored with a 5-point Likert scale. Higher scores represent more powerful beliefs. Total score ranges from 4 to 20
Hospital Anxiety and Depression Scale (HADS) | 1 day
  Hospital Anxiety and Depression Scale (HADS) determines the levels of anxiety and depression that a person is experiencing. The HADS is a fourteen item scale that generates: Seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression.
The Psoriatic Arthritis Quality of Life (PsAQoL) | 1 day
  The Psoriatic Arthritis Quality of Life (PsAQoL) measure is a disease specific patient-reported outcome measure which measures the effect that psoriatic arthritis has on a patient's quality of life. It is a self-administered, 20-item questionnaire that takes about three minutes to complete. The answers are restricted to true or false.A high score on the PsAQoL indicates a lower quality of life. Total score is between 0 and 20.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Fatih, Turkey (Türkiye)

REFERENCES:
- [Background] Hromadkova L, Soukup T, Vlcek J. Quality of life and drug compliance: their interrelationship in rheumatic patients. J Eval Clin Pract. 2015 Oct;21(5):919-24. doi: 10.1111/jep.12399. Epub 2015 Jun 17. PMID 26083391
- [Background] Tolu S, Rezvani A, Karacan I, Bugdayci D, Kucuk HC, Bucak OF, Aydin T. Self-Reported Medication Adherence in Patients With Ankylosing Spondylitis: The Role of Illness Perception and Medication Beliefs. Arch Rheumatol. 2020 Feb 7;35(4):495-505. doi: 10.46497/ArchRheumatol.2020.7732. eCollection 2020 Dec. PMID 33758806